CLINICAL TRIAL: NCT00167687
Title: A Double-Blind Placebo-Controlled Trial of Prazosin for the Treatment of Alcohol Dependence
Brief Title: Prazosin Alcohol Dependence IVR Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Tracy Simpson, Ph.D., Seattle VA Medical Center
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 05-5895-V 02
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Alcoholism
Keywords: Alcoholism; Randomized Controlled Trial
MeSH Terms: conditions — Alcoholism | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Placebo Comparator)
  Interventions: Drug: prazosin

INTERVENTIONS:
Drug: prazosin — Pharmacological treatment: In order to prevent the possible side effect of first-dose hypotension, all participants will receive only 1mg of study medication or placebo nightly for the first two days of study participation. Titration will proceed according to the following schedule:
  Prazosin Dosing: 9 AM 3 PM 9 PM Days 1-2 1 mg (one capsule) Days 3-4 1 mg 1 mg 1 mg Days 5-7 2 mg 2 mg 2 mg Day 8-10 2 mg 2 mg 6 mg Day 11-14 4 mg 4 mg 6 mg Day 15-42 4 mg 4 mg 8 mg

SUMMARY:
This double-blind placebo controlled pilot trial will test the hypothesis that prazosin, an alpha-1 adrenergic receptor antagonist, reduced alcohol consumption and alcohol craving in alcohol dependent individuals without Post Traumatic Stress Disorder (PTSD). The intervention period is six weeks.

DETAILED DESCRIPTION:
The objective of the project is to determine whether prazosin, an alpha-1 adrenergic receptor antagonist, decreases alcohol consumption and/or the subjective experience of alcohol craving in individuals without post-traumatic stress disorder (PTSD) who are seeking treatment for alcohol dependence.

The study hypotheses are: (1) Subjects treated with prazosin will report fewer drinking days and fewer drinks per drinking day than subjects treated with placebo, (2) subjects treated with prazosin will report decreased craving for alcohol as compared to subjects in the placebo condition, and (3) prazosin will be well-tolerated at the proposed dosage by subjects in the prazosin condition compared to subjects in the placebo condition.

This project is a double-blind, randomized, placebo-controlled trial of prazosin in subjects who are dependent on alcohol and have used alcohol within the last 30 days prior to randomization. The treatment phase will last 6 weeks and will include 40 subjects; 20 randomized to each experimental condition (prazosin and placebo). Participants in both the groups will be provided the same behavioral treatment for alcohol dependence throughout the course of the study. Participants in both groups will also use daily Interactive Voice Response (IVR) symptom monitoring technology to track daily fluctuations in alcohol use and craving, as well as medication compliance.

The study will be conducted at the Addiction Treatment Center (ATC) at VAPSHCS, Seattle division.

Participants will include 40 alcohol-dependent adults presenting for chemical dependency treatment at the VA Puget Sound Health Care System (VAPSHCS) Addiction Treatment Center as well as subjects recruited from the general public via advertisements in local weekly newspapers.

Study Procedures: Once potential study participants have undergone an initial screen to insure basic eligibility they will provide informed consent and will undergo a 2-hour baseline assessment that will include completing a diagnostic interview, paper-and-pencil packet of measures, and providing urine and blood specimens. After completion of these assessments, a final determination will be made within three business days as to whether the potential participant meets inclusion but not exclusion criteria. Eligible participants will then be randomized to one of the two treatment groups. The participants will be prompted three times each day by text messaging pages reminding them to take their study medications.

The behavioral treatment to be used in this study is the Medication Management protocol adapted from the procedure used in Project COMBINE. A clinical rescue strategy will be in place such that any participants who evidence severe clinical deterioration including consuming more than 140 standard equivalent drinks in any 7 day period will be removed from the protocol and offered inpatient treatment at VA PSHCS.

During the first two weeks of the study, participants will have twice-weekly orthostatic vital sign and adverse events monitoring by the study nurse or physician, then weekly thereafter. All serious or unexpected adverse events will be reported to the FDA and UW Human Subjects Committee in accordance with requirements. When participants have completed their medication treatment at 6 weeks post-randomization, they will repeat all the baseline measures and laboratory tests (urine and blood samples will be requested) except for the PCL and the California Verbal Learning Test.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years of age or older
* current DSM-IV diagnosis of alcohol dependence with some use in last 30 days
* capacity to provide informed consent
* no planned absences during six week active treatment period that would prevent weekly check-in wiht the study psychiatrist
* English fluency

Exclusion Criteria:

* Score 50 or greater on the PTSD Check List which suggests a current diagnosis of PTSD
* Psychiatric disorder requiring any medication other than anti-depressants
* Current diagnosis of opiate dependence or abuse, chronic treatment with any opiate-containing medications during the previous month, or urine positive for opioids
* Significant acute or chronic medical illness, including unstable angina, recent myocardial infarction, history of congestive heart failure, preexisting hypotension (systolic lower than 110) or orthostatic hypotension (systolic drop greater than 20mmHg after two minutes standing or any drop with dizziness), insulin-dependent diabetes mellitus; chronic renal or hepatic failure, pancreatitis, gout, Meniere's disease, benign positional vertigo, narcolepsy
* Concomitant use of trazodone, tadalafil or verdenafil
* History of prazosin-sensitivity
* Women who are pregnant, nursing infant(s), or of childbearing potential and not using a contraceptive method judged by the investigator to be effective
* Signs or symptoms of alcohol withdrawal at the time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Number of days drinking during the six week intervention | 6 weeks
Number of drinks per drinking day consumed | 6 weeks

SECONDARY OUTCOMES:
Daily craving intensity over the six week intervention | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Simpson, PhD, Principal Investigator — VA Puget Sound Health Care System; Andrew Saxon, MD, Principal Investigator — VA Puget Sound Health Care System; Charles Meredith, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- See also: Interactive Voice Response system vendor — http://www.prosodieinteractive.com/